CLINICAL TRIAL: NCT06671145
Title: Study of New Simple Maneuvers for Differentiating Atrioventricular Nodal Reentry Tachycardia from Orthodromic Atrioventricular Reentry Tachycardia During Electrophysiological Study
Brief Title: Differentiate AVNRT from Orthodromic AVRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam El Din Mohamed Farghaly, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AVNRT and orthodromic AVRT
Record Dates: First submitted 2024-10-20; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: SVT
Keywords: AVNRT - orthodromic AVRT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group (1)catheter ablation after diagnosis of Atrioventricular Nodal Reentry Tachycardia (Active Comparator): diagnosis Atrioventricular Nodal Reentry Tachycardia before catheter ablation
  Interventions: Diagnostic Test: catheter ablation
- group (2) catheter ablation after diagnosis of orthodromic Atrioventricular Reentry Tachycardia (Active Comparator): diagnosis of orthodromic Atrioventricular Reentry Tachycardia before catheter ablation
  Interventions: Diagnostic Test: catheter ablation

INTERVENTIONS:
Diagnostic Test: catheter ablation — Catheter ablation after differentiating Atrioventricular Nodal Reentry Tachycardia from Orthodromic Atrioventricular Reentry Tachycardia during electrophysiological study.

SUMMARY:
To study new maneuvers to differentiate AVNRT from orthodromic AVRT including VA interval variability at tachycardia induction, SA-VA base and local VA index (difference between local VA interval, measured on the coronary sinus catheter during tachycardia and entrainment, at the site of earliest atrial activity).

DETAILED DESCRIPTION:
The differentiation of atrioventricular nodal reentrant tachycardia (AVNRT) from atrioventricular reciprocating tachycardia (AVRT) as well as the localization of accessory pathways (APs) is necessary to guide the catheter ablation of supraventricular tachycardia (SVT). However, existing techniques may prove challenging in differentiating atypical forms of AVNRT from AVRT using a septal AP; or localizing AVRT with different septal AP insertion sites.

There are many diagnostic maneuvers during electrophysiological study eg ventriculo atrial interval (VA) during tachycardia, postpacing interval tachycardia cycle length (PPI-TCL) and stimulus atrial ventriculaoatrial interval (SA-VA). It is important to recognize that as with most diagnostic tests, no single observation or maneuver is 100% sensitive or specific. Therefore, it is important to obtain data from multiple observations and maneuvers to verify the diagnosis.

Also, utility of these techniques usually depends on the tachycardia to be sustained, however sometimes tachycardia is rapidly terminating. VA interval at initiation of tachycardia is usually variable and becomes fixed after several beats. This may be explained by differences in retrograde conduction between AVRT and AVNRT which may be better exposed at the time of tachycardia induction, So measuring the number of beats until VA becomes fixed may theoretically help in differentiating AVNRT from AVRT.

Although several reports have demonstrated the usefulness of the SA-VA using right ventricular (RV) apical stimulation (SA-VAapex) to distinguish AVNRT from AVRT, there remains significant overlap in the SA-VA complicating the distinction between these 2 arrhythmias.

Theoretically, stimulation from the RV basal septum (SA-VAbase) would be expected to shorten the SA interval in AVRT because atrioventricular pathways insert in the ventricular base. On the other hand, the SA-VAbase should have the opposite effect on AVNRT because the impulse must first pass from the RV base to the apex to access the right bundle.

ELIGIBILITY:
Inclusion Criteria:

* All patients with documented narrow complex supraventricular tachycardia presented to electrophysiology lab including all age and sex patients (in Assiut university cath. lab) and proved to be AVNRT or orthodromic AVRT.

Exclusion Criteria:

1. Atrial tachycardia
2. Atrial flutter.
3. Atrial fibrillation.
4. Manifest preexcitation on surface ECG -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
To differentiate between narrow complex supraventricular tachycardia (AVNRT from orthodromic AVRT during electrothysiological study). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Ahmed Fouad, pro, Principal Investigator — Assiut University; Heba Mahmoud Abdel Mohsen El- naggar, Ass. pro, Principal Investigator — Assiut University; marwan sayed mahmoud, doctor, Principal Investigator — Assiut University